CLINICAL TRIAL: NCT04518371
Title: Clinical Performance and Wear Resistance of Milled Resin Composite Material Versus Direct Nanohybrid Bulk-Fill Resin Composite in Restoration of Endodontically Treated Posterior Teeth Over One Year: Randomized Clinical Trial
Brief Title: Clinical Performance of Milled Resin Composite in Restoration of Endodontically Treated Posterior Teeth Over One Year
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Esmeail Hussien, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU-EEHussien
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Endodontically Treated Teeth
Keywords: Endodontically Treated Teeth; Milled Composite; Clinical Performance; Occlusal Wear; IntraOral Scanner
MeSH Terms: conditions — Tooth, Nonvital; Tooth Attrition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect Restoration (Experimental): Milled Resin Composite Block, Shock-absorbing effect due to the dentine-like modulus of elasticity makes BRILLIANT Crios extremely well suited for implant restorations.it is composed of dental glass (barium glass ˂ 1.0 μm), amorphous silica (Sio2 ˂ 20 nm), resin matrix (cross-linked methacrylates) and pigments (inorganic pigments such as ferrous oxide or titanium dioxide).
  Interventions: Other: Reinforced composite for the fabrication of permanent, indirect restorations using a CAD/CAM grinding process.
- Direct Restoration (Active Comparator): 3M™ Filtek™ One Bulk Fill Restorative is a visible light activated, restorative composite optimized to create fast and easy restorations.
  It is composed of fillers which are a combination of a non-agglomerated/non-aggregated 20 nm silica filler, 4 to 11 nm zirconia filler, zirconia/silica cluster filler and ytterbium trifluoride filler consisting of 100nm particles. The inorganic filler loading is about 76.5% by weight (58.5% by volume).
  Interventions: Other: Reinforced composite for the fabrication of permanent, indirect restorations using a CAD/CAM grinding process.

INTERVENTIONS:
Other: Reinforced composite for the fabrication of permanent, indirect restorations using a CAD/CAM grinding process. — Shock-absorbing effect due to the dentine-like modulus of elasticity makes BRILLIANT Crios extremely well suited for implant restorations.it is composed of dental glass (barium glass ˂ 1.0 μm), amorphous silica (Sio2 ˂ 20 nm), resin matrix (cross-linked methacrylates) and pigments
  Other Names: CAD/CAM Composite endo-crown

SUMMARY:
In patients with endodontically treated teeth, will the Indirect Milled composite Endo-crown restorations have a better clinical performance and more wear resistance than the Direct Bulk-Fill resin composite restorations over one year?

Primary Objective: To evaluate clinical performance of different Techniques of Composite Restorations (Indirect restorations using a CAD/CAM grinding process, BRILLIANT Crios, Coltène/Whaledent AG, Switzerland or Direct a light-cured, bulk-fill nanocomposite restorative material, Filtek™ One Bulk Fill Restorative, 3M ESPE Dental Products, USA) in Endodontically treated posterior teeth.

DETAILED DESCRIPTION:
The study will be conducted in Conservative Dentistry Department, Faculty of Dentistry, Cairo University; The operator in charge will be Esraa Esmeail Hussien.

Null-hypothesis: There are no differences in the clinical performance of indirect CAD/CAM milled composite when compared to direct bulk-fil composite endocrowns when in the posterior area.

Aim: This clinical trial will be conducted to assess the clinical performance of using indirect Milled composite or direct bulk-fill resin composite Endo-crowns for restoring the endo-treated teeth, as well to measure the amount of wear on the occlusal tables of both restorations using Digital Scanner.

Patients will be selected from the outpatient clinic of the department Conservative Dentistry Department, Faculty of Dentistry, Cairo University

Clinical Steps:

* A tapered stone with rounded end in a high-speed handpiece with air /water coolant will be used to properly prepare the cavity walls to receive the indirect restoration and any remaining carious dentin will be excavated and removed.
* Cuspal tipping will be done by a wheel stone about 1.5-2mm.
* The entrance to the pulpal canal will be opened. Gutta percha will be removed to a depth not exceeding 2 mm to take advantage of the saddle-like anatomy of the cavity floor. This should be done with a nonabrasive instrument to maintain the integrity of the canal's entrance. No drilling into the dentin will be carried out.
* Any remaining undercuts will be blocked with conventional resin composite.
* The impression will be taken, and the final restoration will be fabricated either direct or indirect.
* The final restoration should be checked intraorally for proximal contacts, occlusion and marginal fit before cementation.
* Isolation of operatory field using rubber dam.
* Selective enamel etching technique will be applied for bonding of tooth structure, 35-40% phosphoric acid gel will be applied to the enamel margins only for 15 seconds, rinsed for 15 seconds and gently dried by cotton pellet.
* Adhesive will be used according to the manufacturers' instructions.
* Adhesive resin cement will be applied into the preparation. The restoration will be placed in the cavity and checked for complete seating. The cement will be light cured for only 2 seconds to facilitate removal of the excess. Then light curing will be done from all directions each for 40 seconds for achieving the final set.
* The proximal contacts will be checked with dental floss.
* The occlusion will be adjusted using articulating paper.
* Finishing and Polishing using finishing stones and polishing rubber points.

Primary Objective: To evaluate clinical performance of different Techniques of Composite Restorations (Indirect restorations using a CAD/CAM grinding process, BRILLIANT Crios, Coltène/Whaledent AG, Switzerland or Direct a light-cured, bulk-fill nanocomposite restorative material, Filtek™ One Bulk Fill Restorative, 3M ESPE Dental Products, USA) in Endodontically treated posterior teeth.

ELIGIBILITY:
Inclusion Criteria of participants:

* Patients with asymptomatic endodontically treated molars.
* Males or Females.
* Good oral hygiene.
* Co-operative patients approving to participate in the study.

Inclusion Criteria of teeth:

* Asymptomatic endodontically treated upper or lower molars with
* Homogenous root canal filling ending 1-2mm from the radiographic apex.
* Proximal compound cavities.
* Favorable occlusion.

Exclusion criteria of participants:

* High caries index with poor oral hygiene.
* Severe medical complications.
* Pregnancy.
* Allergic history concerning methacrylates Disabilities.
* Heavy smoking.
* Xerostomia.
* Lack of compliance.
* Evidence of parafunctional habits.
* Temporomandibular joint disorders.

Exclusion criteria of the teeth:

* Teeth with remaining wall thickness less than 1mm.
* Teeth with improper or symptomatic endodontic treatment.
* Deep subgingival cavity margins.
* Possible future prosthodontic restoration of teeth.
* Severe periodontal problems.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Degree of Continuity between natural tooth structure and the restoration | Immediately after procedure
  Tactile sensation checking the anatomic form to show if there is no discontinuity, Slight discontinuity, or discontinuity and failure
Degree of Continuity between natural tooth structure and the restoration | 6 months
  Tactile sensation checking the anatomic form to show if there is no discontinuity, Slight discontinuity, or discontinuity and failure
Degree of Continuity between natural tooth structure and the restoration | 12 months
  Tactile sensation checking the anatomic form to show if there is no discontinuity, Slight discontinuity, or discontinuity and failure

SECONDARY OUTCOMES:
The degree of mismatch from the normal range of tooth shades and translucency | Immediately after procedure
  Visual inspection to check the proximity of the shade from the natural tooth
The degree of mismatch from the normal range of tooth shades and translucency | 6 months
  Visual inspection to check the proximity of the shade from the natural tooth
The degree of mismatch from the normal range of tooth shades and translucency | 12 months
  Visual inspection to check the proximity of the shade from the natural tooth
Distance penetrated due to secondary caries by visual evidence of dark keep discoloration adjacent to the restoration but not directly associated with cavosurface margins | Immediately after procedure
  Visual inspection of discoloration that occurs on the tooth after the filling has been used for a period of time
Distance penetrated due to secondary caries by visual evidence of dark keep discoloration adjacent to the restoration but not directly associated with cavosurface margins | 6 months
  Visual inspection of discoloration that occurs on the tooth after the filling has been used for a period of time
Distance penetrated due to secondary caries by visual evidence of dark keep discoloration adjacent to the restoration but not directly associated with cavosurface margins | 12 months
  Visual inspection of discoloration that occurs on the tooth after the filling has been used for a period of time
Pain due to dentin hypersensitivity (evaporative stimulus) | Immediately after procedure
  Pain arising from dentin hypersensitivity around the restoration stimulated by air blast measured by YES or NO scale
Pain due to dentin hypersensitivity (evaporative stimulus) | 6 months
  Pain arising from dentin hypersensitivity around the restoration stimulated by air blast measured by YES or NO scale
Pain due to dentin hypersensitivity (evaporative stimulus) | 12 months
  Pain arising from dentin hypersensitivity around the restoration stimulated by air blast measured by YES or NO scale
Area of continuous movement of an explorer across the surface of the restoration | Immediately after procedure
  Surface texture is highly polished or gritty containing supramicron-sized particles or Surface pitting is coarse to inhibit the continuous movement of an explorer across the surface
Area of continuous movement of an explorer across the surface of the restoration | 6 months
  Surface texture is highly polished or gritty containing supramicron-sized particles or Surface pitting is coarse to inhibit the continuous movement of an explorer across the surface
Area of continuous movement of an explorer across the surface of the restoration | 12 months
  Surface texture is highly polished or gritty containing supramicron-sized particles or Surface pitting is coarse to inhibit the continuous movement of an explorer across the surface
Distance penetrated by the Explorer at the tooth restoration interface | Immediately after procedure
  The explorer will be drawn across the surface of the restoration toward the tooth
Distance penetrated by the Explorer at the tooth restoration interface | 6 months
  The explorer will be drawn across the surface of the restoration toward the tooth
Distance penetrated by the Explorer at the tooth restoration interface | 12 months
  The explorer will be drawn across the surface of the restoration toward the tooth

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Es Hussien, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt